CLINICAL TRIAL: NCT02860403
Title: Motor Imagery for Reach-to-grasp Rehabilitation After Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-541
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-08

CONDITIONS: Tetraplegia C5-C6; Tetraplegia C6-C7
Keywords: Cervical spinal cord injury; Motor imagery; Magnetoencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- C6-C7 patients (Experimental): C6-C7 patients able to recover tenodesis grasp.
  Interventions: Procedure: motor imagery
- C5-C6 patients (Experimental): C5-C6 patients for whom surgery for rehabilitation of an upper limb is indicated with a upper limit of one year after trauma, and after complete clinical and functional evaluation
  Interventions: Procedure: motor imagery
- Control group (No Intervention): a control group (n=6) matched on age and sex to C6-C7 without medical history or neurological disorder

INTERVENTIONS:
Procedure: motor imagery — Intervention consisted of supervised MI during which the participants were trained to imagine performing a single-joint wrist extension movement and a multiple-joint reach-to-grasp movement using tenodesis. The two movements were practiced in separate blocks and each 45 minute MI session consisted of six to eight blocks. Within a given block patients; i) performed the movement once, ii) imagined it using visual imagery (between five and ten repetitions), iii) performed the movement again, and iv) imagined it using kinesthetic imagery (between five and ten repetitions). All movements (performed and imagined) were timed by the experimenter to ensure that the durations of both imagined and physically practiced movements were similar. Imagery vividness was controlled with self-rated assessments using a visual analogic scale (from 0, the image or feeling was absent, to 10 when it was as clear or intense as physical practice).
  Arms: C5-C6 patients; C6-C7 patients

SUMMARY:
Single center, pilot study, to evaluate the influence of Motor Imagery (MI) on functional rehabilitation and cerebral plasticity through the qualitative and quantitative mental practice approach. For this, the investigators will use magnetoencephalography (MEG) but also physiological and behavioral indicators developed by the Laboratoire de la Performance Motrice, Mentale et du Matériel (P3M) of Université Claude Bernard Lyon 1 and its partners.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old,
* quadriplegia elicited by spinal cord injury (SCI) at the C5, C5-C6, C6, or C6-C7 level,
* complete infra-lesional motor deficit according to the ASIA impairment scale with finger and forearm flexor muscles paralysis,
* post-traumatic period >6 months (since a motor recovery plateau is usually reached at 6-month post-SCI

Exclusion Criteria:

* non-stabilized hypertension or pathological autonomic nervous system dysfunction (e.g., orthostatic hypotension),
* cerebral damage and/or cognitive deficit,
* elbow or shoulder joint amplitude restriction, upper limb para-osteoarthropathy,
* participation to another study
* presence of metallic objects within the body incompatible with MEG or functional magnetic resonance imaging (fMRI) recordings.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Motor imagery ability | 10 weeks
  Motor imagery ability assessed by magnetoencephalography measurements

SECONDARY OUTCOMES:
Movement time (MT) | 10 weeks
  Kinematic parameters of movement: temporal parameters: movement time (MT)
absolute time to peak velocity | 10 weeks
  Kinematic parameters of movement: temporal parameters: absolute time to peak velocity
movement amplitude at peak velocity | 10 weeks
  Kinematic parameters of movement: temporal parameters: movement amplitude at peak velocity
time to opening | 10 weeks
  Kinematic parameters of movement: temporal parameters: time to opening
time to maximal opening | 10 weeks
  Kinematic parameters of movement: temporal parameters: time to maximal opening
amplitude of maximal opening | 10 weeks
  Kinematic parameters of movement: temporal parameters: amplitude of maximal opening
Trajectory of movement measured in the XY plane | 10 weeks
  Kinematic parameters of movement: spatial parameters: Trajectory of movement measured in the XY plane
height of elbow and wrist at the moment of grasping an object, measured in mm in the YZ plane | 10 weeks
  Kinematic parameters of movement: spatial parameters: height of elbow and wrist at the moment of grasping an object, measured in mm in the YZ plane
muscular force evaluated by muscle testing performed by a physiotherapist | 10 weeks
  muscular force evaluated by muscle testing performed by a physiotherapist (score from 0 to 5)
joint amplitude evaluated in degrees (°) by the physiotherapist | 10 weeks
Box and Block test | 10 weeks
  Box and Block test performed by an occupational therapist
Minnesota test. | 10 weeks
  Minnesota test performed by an occupational therapist
amplitude of electrodermal responses | 10 weeks
  mental chronometric assessment associated with acquisition of electrodermal responses
duration of electrodermal responses | 10 weeks
  mental chronometric assessment associated with acquisition of electrodermal responses
Kinesthetic and Visual Imagery Questionnaire | 10 weeks
  The Kinesthetic and Visual Imagery Questionnaire (KVIQ) will allow a qualitative evaluation of the mental representation capacity of patients

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RODE, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Henry Gabrielle - Médecine physique et Réadaptation, Hospices Civils de Lyon, 20 Route de Vourles,, Saint-Genis-Laval, France

REFERENCES:
- [Result] Mateo S, Reilly KT, Collet C, Rode G. Descriptive pilot study of vividness and temporal equivalence during motor imagery training after quadriplegia. Ann Phys Rehabil Med. 2018 Sep;61(5):300-308. doi: 10.1016/j.rehab.2018.06.003. Epub 2018 Jun 23. PMID 29944923